CLINICAL TRIAL: NCT00319670
Title: A Pilot Study of a New MiraLax® Dose Formulation For Use in Constipated Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 851-201
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Constipation
Keywords: constipation; pediatric
MeSH Terms: conditions — Constipation | interventions — polyethylene glycol 3350

INTERVENTIONS:
Drug: MiraLax

SUMMARY:
To evaluate patient acceptance of a new MiraLax dose formulation in children currently treated with polyethylene glycol 3350 powder for treatment of constipation.

DETAILED DESCRIPTION:
To evaluate patient acceptance of a new MiraLax dose formulation in children currently treated with polyethylene glycol 3350 powder for treatment of constipation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female constipated outpatients between the ages of 4 and 16
2. Currently taking a dose of less than or equal to 17g of PEG 3350 powder that has been consistent for at least 4 weeks
3. Current treatment is considered successful - defined as greater than 2 bowel movements per week with no accidents
4. Are otherwise in good health, as judged by a physical examination
5. If female and of childbearing potential, patient must be using oral contraceptives, depot contraceptives, intrauterine device, or testifies that she is monogamous with a vasectomized partner, or practices abstinence and will continue to do so during the duration of study
6. In the investigator's judgment, patient or guardian is mentally competent to sign an instrument of informed consent

Exclusion Criteria:

1. Patients with heme positive stool at baseline exam
2. Patients who are impacted at baseline exam
3. Patients that are not receiving PEG 3350
4. Patients on PEG 3350 that continue to have problems
5. Patients with known or suspected perforation or obstruction
6. Patients with a history of gastric retention, inflammatory bowel disease, bowel resection, or colostomy
7. Patients with a known history of organic cause for their constipation.
8. Patients currently using medications known to cause constipation. These include Opiates, antidepressants, SSRI's, antimotility agents and anticholinergics.
9. Patients who are breastfeeding, pregnant, or intend to become pregnant during the study
10. Female patients of childbearing potential who refuse a pregnancy test
11. Patients who, in the opinion of the investigator, should not be included in the study for any reason, including inability to follow study procedure
12. Patients with known allergy to PEG or PEG containing medications
13. Patients who, within the past 30 days have participated in an investigational clinical study

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25
Dates: Start 2006-03; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Efficacy will be measured by analysis of patient self-reported BM data.
Adverse events will be monitored and analyzed for safety purposes.

SECONDARY OUTCOMES:
Patient acceptance will be measured by analysis of subjective questionnaire data.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Nurko, MD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Boston, Massachusetts
  - Youngstown, Ohio